CLINICAL TRIAL: NCT07173400
Title: Effects of Transcutaneous Auricular Vagus Nerve Stimulation on Symptom Severity, Sleep Quality, Central Sensitization, and Kinesiophobia in Fibromyalgia: A Randomized Controlled Trial
Brief Title: Effects of Transcutaneous Auricular Vagus Nerve Stimulation on Symptom Severity, Sleep Quality, Central Sensitization, and Kinesiophobia in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hatice Betigul Meral (Other)
Responsible Party: Sponsor-Investigator, Hatice Betigul Meral, Principal Investigator, Medipol University
Organization: Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-4945 (30/0
Record Dates: First submitted 2025-09-05; First posted 2025-09-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia (FM); Chronic Pain
Keywords: Vagal Nerve Stimulation; fibromyalgia; pain; chronic pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Pain

STUDY DESIGN:
Intervention Model Description: This study used a two-arm, randomized, sham-controlled, parallel group design with a 1:1 allocation ratio
Who Masked: Participant
Masking Description: Participants and outcome assessors were blinded to group allocation. The treating clinician who applied stimulation was aware of assignment but did not participate in outcome assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TaVNS (Experimental): Participants received active transcutaneous auricular vagus nerve stimulation (TaVNS) using the VagusStim® device (Vagus Medical Technologies, Istanbul, Türkiye). The electrode was placed on the left cymba concha and stimulation was applied for 30 minutes per day, 5 days per week, over 4 weeks (20 sessions). Stimulation parameters included 1-30 Hz frequency, 50-250 μs pulse width, and current individually adjusted (0.1-36 mA) to each participant's sensory threshold.
  Interventions: Device: Active Transcutaneous Auricular Vagus Nerve Stimulation (TaVNS)
- Sham TaVNS (Placebo Comparator): Participants underwent sham stimulation using the same VagusStim® device under identical conditions. The electrode was placed on the left earlobe, an area without vagal innervation, and sessions lasted 30 minutes per day, 5 days per week, for 4 weeks. No effective vagus nerve stimulation was delivered, maintaining participant blinding.
  Interventions: Device: Sham Transcutaneous Auricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Active Transcutaneous Auricular Vagus Nerve Stimulation (TaVNS) — Active TaVNS delivered with the VagusStim® device (Vagus Medical Technologies, Istanbul, Türkiye). The bipolar electrode was placed on the left cymba concha. Stimulation was applied for 30 minutes per day, 5 days per week, for 4 weeks (20 sessions). Parameters included frequency 1-30 Hz, pulse width 50-250 μs, and current intensity individually adjusted (0.1-36 mA) to the participant's sensory threshold.
  Arms: Active TaVNS
Device: Sham Transcutaneous Auricular Vagus Nerve Stimulation — Sham stimulation delivered with the same VagusStim® device under identical conditions. The electrode was rotated and placed on the left earlobe, which lacks vagal innervation. Sessions lasted 30 minutes per day, 5 days per week, for 4 weeks (20 sessions). No effective vagus nerve stimulation was delivered, preserving participant blinding.
  Arms: Sham TaVNS

SUMMARY:
Fibromyalgia is a chronic condition characterized by widespread musculoskeletal pain, fatigue, sleep disturbances, and sensitivity to touch. Current treatments often provide only partial relief. This study evaluates a non-invasive technique called transcutaneous auricular vagus nerve stimulation (TaVNS), which delivers gentle electrical impulses to a part of the ear connected to the vagus nerve. The vagus nerve plays an important role in regulating pain, stress, and autonomic body functions such as sleep.

In this randomized controlled pilot trial, participants with fibromyalgia are assigned to receive either active TaVNS or sham (placebo) stimulation for 30 minutes per day, five days per week, over a four-week period. Participants are followed for a total of 8 weeks. The investigators will assess outcomes including pain intensity, sleep quality, central sensitization, and fear of movement (kinesiophobia).

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic pain syndrome associated with widespread musculoskeletal pain, fatigue, sleep disturbances, and autonomic dysregulation. Current treatments provide only partial relief, highlighting the need for novel therapeutic approaches.

Rationale:

The vagus nerve is a key regulator of autonomic and inflammatory processes. Transcutaneous auricular vagus nerve stimulation (TaVNS) is a non-invasive technique that can modulate vagal activity through electrodes placed on the external ear, offering a potential alternative to surgically implanted vagus nerve stimulators.

Study Design:

This is a randomized, sham-controlled pilot trial conducted at Istanbul Medipol University. Thirty participants with fibromyalgia are randomized in a 1:1 ratio to receive either active TaVNS or sham stimulation.

Intervention:

Device: VagusStim® (Vagus Medical Technologies, Istanbul, Türkiye; CE-marked).

Electrode placement: left cymba concha (active group) vs. left earlobe (sham group).

Stimulation parameters: frequency 1-30 Hz, pulse width 50-250 μs, current intensity individually adjusted (0.1-36 mA) to each participant's sensory threshold.

Schedule: 30 minutes per day, 5 days per week, for 4 consecutive weeks (20 sessions total).

Supervision: All sessions are clinician-supervised.

Outcome Measures:

Primary outcomes:

Pittsburgh Sleep Quality Index (PSQI) - subjective sleep quality.

Fibromyalgia Impact Questionnaire (FIQ) - disease severity and functional impact.

Central Sensitization Inventory (CSI) - symptoms related to central sensitization.

Secondary outcomes:

Visual Analog Scale (VAS) - pain intensity.

Tampa Scale for Kinesiophobia (TSK) - fear of movement.

Symptom Severity Scale (SSS).

Widespread Pain Index (WPI).

Assessment timepoints: baseline, week 2, week 4, and week 8.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 65 years

Diagnosis of fibromyalgia according to the 2016 revised ACR criteria

Receiving stable pharmacological and/or non-pharmacological treatment for at least 3 months

Ability to understand study procedures and provide informed consent

Exclusion Criteria:

Pregnancy

History of epilepsy or cardiac arrhythmia

Acute or chronic infection

Heart failure (NYHA class II-IV)

Renal failure stage II or higher

Active malignancy

Psychotic disorders or current psychiatric treatment

Diagnosis of immune-mediated rheumatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | Baseline, Week 2, Week 4, Week 8
  The FIQ evaluates the overall health status and functional impact of fibromyalgia, including physical functioning, pain, fatigue, and mood. Scores range from 0 to 100, with higher scores reflecting greater disease impact.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, Week 2, Week 4, Week 8
  The PSQI is a validated self-report questionnaire that assesses subjective sleep quality and disturbances over the past month. Scores range from 0 to 21, with higher scores indicating poorer sleep quality.
Central Sensitization Inventory (CSI) | Baseline, Week 2, Week 4, Week 8
  The CSI is a 25-item self-report questionnaire assessing symptoms related to central sensitization, including sensitivity to pain, fatigue, and cognitive complaints. Scores range from 0 to 100, with higher scores indicating greater sensitization.

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia (TSK) | Baseline, Week 2, Week 4, Week 8
  The TSK is a 17-item self-report questionnaire measuring fear of movement or reinjury. Items are scored on a 4-point Likert scale, with total scores ranging from 17 to 68. Higher scores indicate greater kinesiophobia.
Visual Analog Scale (VAS) for Pain | Baseline, Week 2, Week 4, Week 8
  Pain intensity is assessed using a 10-cm visual analog scale, with 0 representing "no pain" and 10 representing "worst imaginable pain." Participants mark their pain level along the line, which is recorded as a numeric score.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Bagcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study is a small, single-center pilot trial. Due to the limited sample size and ethical/privacy considerations, individual participant data will not be shared in a public repository. De-identified data may be made available from the corresponding author upon reasonable request.

REFERENCES:
- [Result] Paccione CE, Stubhaug A, Diep LM, Rosseland LA, Jacobsen HB. Meditative-based diaphragmatic breathing vs. vagus nerve stimulation in the treatment of fibromyalgia-A randomized controlled trial: Body vs. machine. Front Neurol. 2022 Nov 3;13:1030927. doi: 10.3389/fneur.2022.1030927. eCollection 2022. PMID 36438970
- [Result] Abdel-Baset AM, Abdellatif MA, Ahmed HHS, El Shaarawy NK. Pain neuroscience education versus transcutaneous vagal nerve stimulation in the management of patients with fibromyalgia. Egypt Rheumatol. 2023;45:191-195. doi:10.1016/j.ejr.2023.03.001.
- [Result] Kutlu N, Ozden AV, Alptekin HK, Alptekin JO. The Impact of Auricular Vagus Nerve Stimulation on Pain and Life Quality in Patients with Fibromyalgia Syndrome. Biomed Res Int. 2020 Feb 28;2020:8656218. doi: 10.1155/2020/8656218. eCollection 2020. PMID 32190684
- [Result] Turk Kalkan T, Tarakci D, Kilic G, Celikyurt C. Investigation of the Effectiveness of Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) and Vestibular Rehabilitation in Patients with Unilateral Vestibular Hypofunction. Medicina (Kaunas). 2025 May 9;61(5):872. doi: 10.3390/medicina61050872. PMID 40428830